CLINICAL TRIAL: NCT04216420
Title: Electronic Pillbox-enabled Self-administered Therapy Versus Standard Directly Observed Therapy for Tuberculosis Medication Adherence and Treatment Outcomes in Ethiopia: a Multicenter Randomized Controlled Trial
Brief Title: Electronic Pillbox-enabled SAT Versus DOT for TB Medication Adherence and Treatment Outcomes
Acronym: SELFTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Collaborators: Emory University School of Medicine, US (Unknown); Armauer Hansen Research Institute, Ethiopia (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Dr. Tsegahun Manyazewal, Principal Investigator, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 077/19/CDT; D43TW009127 (NIH)
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Medication event reminder monitor; Self-administered therapy; Directly observed therapy (DOT); Adherence; Treatement outcome; Digital health; Ethiopia
MeSH Terms: conditions — Tuberculosis; Directly Observed Therapy

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, controlled, open-label, non-inferiority, effectiveness-implementation type 2 hybrid trial.
Who Masked: Outcomes Assessor
Masking Description: Permuted block randomization method was used to randomly allocate participants and maintain a balance of the number of participants assigned to each arm. The study investigators who were responsible for assessing study outcomes and writing the report were blinded to group allocation until the manuscript was completed. A statistician masked to group allocation performed the analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MERM-observed self-administered therapy (SAT) (Experimental): A participant in the intervention arm (n = 57) will receive a 15-day TB medication supply in the evriMED500 MERM device to self-administer. The participant returns every 15 days, where the healthcare provider counts any remaining tablets in the pillbox device, connects the MERM module with a computer and downloads the pill-taking data, reviews the event reports together with the participant and captures the data, underwent IsoScreen urine isoniazid test and refills the participant with a 15-day medication supply in the MERM device.
  Interventions: Device: MERM-observed self-administered therapy
- Standard directly observed therapy (DOT) (No Intervention): The provider handles a participant in the control arm (n = 57) according to the standard DOT, where the participant visits the healthcare facility each day throughout the intensive phase to swallow the daily dose with direct observation by the healthcare provider. The participant will undergo the urine isoniazid test every 15 days.
  Both arms will be treated based on the WHO-recommended two-month fixed-dose-combination of first-line anti-TB drug (2RHZE) delivered as a single daily dose and followed throughout the intensive phase that lasts two months. In the end, participants will undergo a microbiological test to assess sputum smear conversion and trained study staff will complete several data tools, including a treatment outcome monitoring tool, adherence self-report, HRQoL, cost, treatment satisfaction, and MERM usability tools.

INTERVENTIONS:
Device: MERM-observed self-administered therapy — The MERM device has an electronic module and a medication container that records adherence, stores medication, emits audible and visual on-board alarms to remind patients to take their medications on time and refill, and enables providers to download the data and monitor adherence. It is manufactured by Wisepill Technologies, South Africa.
  Other Names: EvriMed500 medication event reminder monitor
  Arms: MERM-observed self-administered therapy (SAT)

SUMMARY:
To address the multifaceted challenges associated with tuberculosis (TB) in-person directly observed therapy (DOT), the World Health Organization recently recommended countries maximize the use of digital adherence technologies. Sub-Saharan Africa needs to investigate the effectiveness of such technologies in local contexts and proactively contribute to global decisions around patient-centered TB care. This study aims to evaluate the effectiveness of pillbox-enabled self-administered therapy (SAT) compared to standard DOT on adherence to TB medication and treatment outcomes in Ethiopia. It also aims to assess the usability, acceptability, and cost-effectiveness (health-related quality of life and catastrophic costs) of the intervention from the patient and provider perspectives. It is designed as a multicenter, randomized, controlled, open-label, non-inferiority, effectiveness-implementation hybrid, mixed-methods, two-arm trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new or previously treated bacteriologically confirmed drug-sensitive pulmonary TB
* Eligible to start the standard 6-month first-line anti-TB medication
* Outpatient
* Men or women age 18 years and above
* Able and willing to provide informed consent

Exclusion Criteria:

* Patients with known drug-resistant TB
* Any condition that causes cognitive impairment such as severe acute illness or injury, developmental retardation, or severe psychiatric illness and thus precludes informed consent or safely participating in the study procedures
* Inpatients
* Concurrent extrapulmonary TB
* Contraindicated medications
* Active liver disease that requires a TB regimen other than HREZ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Level of adherence | Two months
  Individual-level percentage adherence over the two-month intensive phase measured by adherence records compiled from MERM device vs. DOT records.
Sputum conversion | Before and after the two-month intensive phase
  Participant with sputum smear converted following the standard two-month intensive phase treatment

SECONDARY OUTCOMES:
Negative IsoScreen urine isoniazid test | Two months
  Number of participants with negative IsoScreen urine isoniazid test
Adverse treatment outcome | Two months
  Participants having at least one of the three events: treatment not completed; death; or loss to follow-up.
Self-reported adherence | Two months
  Participants who self-reported to have forgotten to take their medication
Health-related quality of life (HRQoL) | Two months
  The association between MERM-observed therapy and HRQoL, with the HRQoL measured and calculated for each participant by arm using the EuroQoL 5-dimension 5-level (EQ-5D-5L) score ranging from 0 to 1, with a higher score designating better HRQoL.
Catastrophic costs | Two months
  Participants with overall TB treatment cost exceeding or equivalent to 20% of their income.
Post-diagnostic cost from an individual patient's perspective | Two months
  Participant's cumulative direct costs (out-of-pocket costs related to anti-TB drug pick-up) and indirect costs (guardian and coping costs) over the two-month intensive phase.
Patient-reported treatment satisfaction | Two months
  Participant's treatment satisfaction measured using the treatment satisfaction questionnaire for medication version 1.4 (TSQM v1.4) tool on a scale 0 to 100, with higher score indicating better satisfaction.
Patient-reported usability of the MERM device | Two months
  Participant's experience using the MERM device measured by an 18-item questionnaire and the score transformed in to a scale from 0 to 100, with higher score indicating better usability (Intervention arm only).

CONTACTS AND LOCATIONS:
Overall Officials: Henry M Blumberg, MD, Study Director — Emory University School of Medicine and Rollins School of Public Health
Locations (1):
- Addis Ababa University, College of Health Sciences, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Manyazewal T, Woldeamanuel Y, Getinet T, Hoover A, Bobosha K, Fuad O, Getahun B, Fekadu A, Holland DP, Marconi VC. Patient-reported usability and satisfaction with electronic medication event reminder and monitor device for tuberculosis: a multicentre, randomised controlled trial. EClinicalMedicine. 2023 Jan 17;56:101820. doi: 10.1016/j.eclinm.2022.101820. eCollection 2023 Feb. PMID 36684395
- [Derived] Manyazewal T, Woldeamanuel Y, Holland DP, Fekadu A, Marconi VC. Effectiveness of a digital medication event reminder and monitor device for patients with tuberculosis (SELFTB): a multicenter randomized controlled trial. BMC Med. 2022 Sep 28;20(1):310. doi: 10.1186/s12916-022-02521-y. PMID 36167528
- [Derived] Manyazewal T, Woldeamanuel Y, Fekadu A, Holland DP, Marconi VC. Effect of Digital Medication Event Reminder and Monitor-Observed Therapy vs Standard Directly Observed Therapy on Health-Related Quality of Life and Catastrophic Costs in Patients With Tuberculosis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 15;5(9):e2230509. doi: 10.1001/jamanetworkopen.2022.30509. PMID 36107429
- [Derived] Manyazewal T, Woldeamanuel Y, Blumberg HM, Fekadu A, Marconi VC. The potential use of digital health technologies in the African context: a systematic review of evidence from Ethiopia. NPJ Digit Med. 2021 Aug 17;4(1):125. doi: 10.1038/s41746-021-00487-4. PMID 34404895
- [Derived] Manyazewal T, Woldeamanuel Y, Holland DP, Fekadu A, Blumberg HM, Marconi VC. Electronic pillbox-enabled self-administered therapy versus standard directly observed therapy for tuberculosis medication adherence and treatment outcomes in Ethiopia (SELFTB): protocol for a multicenter randomized controlled trial. Trials. 2020 May 5;21(1):383. doi: 10.1186/s13063-020-04324-z. PMID 32370774